CLINICAL TRIAL: NCT06158685
Title: The Effect of Hyperextension Exercises on Pain, Disability, Flexibility and Performance Level in Patients With Lumbar Disc Herniation
Brief Title: The Effect of Hyperextension Exercises In Lumbal Disc Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet GÖĞREMİŞ (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Sponsor-Investigator, Mehmet GÖĞREMİŞ, The Effect of Hyperextension Exercises on Pain, Disability, Flexibility and Performance Level in Patients With Lumbar Disc Herniation, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fztmehmetgogremis123
Record Dates: First submitted 2023-08-03; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Female Patients Diagnosed With LDH at L4-S1
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The control group subjects were applied with 15 sessions of conventional physiotherapy consisting of hotpack, ultrasound, and TENS.
  Interventions: Other: Control Group
- study group (Experimental): The study group subjects received 15 sessions of McKenzie hyperextension exercises in addition to the conventional physiotherapy program.
  Interventions: Other: Study Group

INTERVENTIONS:
Other: Study Group — Treatment: Hyperextension exercises as described by McKenzie (in addition to the conventional physiotherapy program)
  McKenzie Hyperextension Exercises:
  * Exercises:
    1. Prone position, arms by the side, deep breath, relax back muscles, holding for 2-3 minutes.
    2. Prone position, raise trunk by raising head above forearms, elbows at shoulder level, maintaining for 2-3 minutes (10 repetitions).
    3. Prone position, hands at elbow level, straighten elbows, raise the upper body from the floor and backwards as far as pain permits, holding for 2-3 seconds (10 repetitions).
    4. Standing with feet shoulder-width apart, hands on waist, leaning backwards as far as possible from the lumbar region without bending knees, holding for 2-3 seconds (10 repetitions).
       Additional Information:
  * Researcher Consistency: All treatments and evaluations were performed by the same researcher.
  Frequency: 5 days a week Duration: 3 consecutive weeks
  Arms: study group
Other: Control Group — Treatment: Conventional physiotherapy program
  * Components:
    * Hot pack was applied to the lumbar region for 20 minutes
    * Ultrasound (ITO device) at 1 MHz and 1.5 W/cm2 for 5 minutes
    * Transcutaneous Electrical Nerve Stimulation (TENS) at 50-100 Hz for 20 minutes
    * Researcher Consistency: All treatments and evaluations for both groups were performed by the same researcher.
  * Session Duration: An average of 45 minutes per session
  * Frequency: 5 days a week
  * Duration: 3 consecutive weeks
  * Total Sessions: 15
  Arms: control group

SUMMARY:
The aim of this study was to examine the short-term effect on pain severity, disability level, flexibility and performance level of McKenzie hyperextension exercises applied in addition to conventional physiotherapy approaches in patients diagnosed with LDH.

A total of 48 consecutive female patients diagnosed with LDH at L4-S1 were randomly separated into 2 groups of 24 as the study group and control group. The control group subjects were applied with 15 sessions of conventional physiotherapy consisting of hotpack, ultrasound, and TENS. The study group subjects received 15 sessions of McKenzie hyperextension exercises in addition to the conventional physiotherapy program.

DETAILED DESCRIPTION:
Aim: The aim of this study was to examine the short-term effect on pain severity, disability level, flexibility and performance level of McKenzie hyperextension exercises applied in addition to conventional physiotherapy approaches in patients diagnosed with LDH.

Method: A total of 48 consecutive female patients diagnosed with LDH at L4-S1 were randomly separated into 2 groups of 24 as the study group and control group. The control group subjects were applied with 15 sessions of conventional physiotherapy consisting of hotpack, ultrasound, and TENS. The study group subjects received 15 sessions of McKenzie hyperextension exercises in addition to the conventional physiotherapy program. Before treatment, immediately after treatment, and at 3 months after the end of treatment, the two groups were compared in respect of pain severity (Visual Analog Scale- VAS), performance level (Half-Squat Test and The 5 Times Sit-Stand Test), flexibility level (Modified Sit And Reach Test), and disability level (Oswestry Disability Index - ODI).

ELIGIBILITY:
Inclusion Criteria:

* The patients included were diagnosed on MRI with L4-S1 LDH (bulging level),
* were taking no drugs other than simple painkillers,
* had LDH symptoms ongoing for at least 3 months.

Exclusion Criteria:

* Patients were excluded from the study if they had a history of lumbar spinal surgery,
* had any disease involving the lumbar spine other than LDH (piriformis syndrome, infection, spondylosis, spondylolysis, spondylolisthesis, ankylosing spondylitis, spinal stenosis, facet syndrome, spinal malignancy, osteoporosis),
* severe neurological loss,
* diabetes mellitus, or were pregnant.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline and week 8
  This is a simple, reliable and valid scale, used as the most apropriate tool to define the severity and intensity of pain. The VAS is a 10 cm horizontal scale marked from 0-10, where 0= no pain and 10= the most intolerable pain. Subjects are instructed to mark the point on the scale representing the severity of the pain they feel. The marked points were measured and recorded.
Flexibility Evaluation | Baseline and week 8
  To evaluate lumbar region flexibility, The Modified Sit And Reach Test (Back-saver Sit-and-Reach Test - BSRT) was used. This test is applied on a test table 60 cm long, 45cm wide, and 32 cm high, with the subject seated with the legs extended in front. The sole of the foot on the side to be tested rests against the test board with the knee in full extension and the contralateral leg is positioned with the knee in 45-90° flexion and the hip joint in 45° flexion. The subject is then instructed to reach over the test board while in this position. Two plastic measures marked in 1 mm gradations are attached to the board, taking the point where it rests against the foot as zero and extending back by 20 cm and forward by 40 cm. Scores of the reach of the subject were recorded as negative (-) if before the zero point and as positive (+) if after.
Performance Evaluation | Baseline and week 8
  The first test applied to determine the performance level of the subjects was the Half-Squat Test (HST). Throughout 1 minute, the subject is instructed to stand up straight then with the knees in 20° flexion to squat and then return to the upright position. A chronometer was started on the "start" command and at the end of 1 min, the score was recorded of the number of squats performed.
  The second performance test was the 5 x Sit To Stand Test (5x SST). On the "start" command, the subject sits and stands from a chair 5 times. The time was recorded on a chronometer.
Disability Level Evaluation | Baseline and week 8
  The ODI was used to determine the level of disability. The ODI is a scale used to determine the degree of functional incapacity in daily living activities caused by lower back pain. The total score ranges from 0 to 50, with higher points showinga higher level of disability. The points are evaluated as 0-10 points: low level disability, 11-30 points: moderate level disability, 31-50: severe level disability.17 Validity and reliability studies of the Turkish version of the scale were made by Yakut et al.

CONTACTS AND LOCATIONS:
Overall Officials: Ejder Berk, Study Chair — Kahmanamaras Sutcü İmam University
Locations (1):
- KahramanmarasISU, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No